CLINICAL TRIAL: NCT05985824
Title: Comparison of the Effect on the Quality of Life of Lung Cancer Patients Who Underwent Prnayama Breathing Exercise and Did Not Apply Any Exercise.
Brief Title: The Effect of Pranayama Breathing Exercise on Quality of Life in Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Zeynep Doğan, Lecturer, Sanko University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SANKOU-HEM-ZD-01
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Pranayama; Quality of Life; Nursing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with primary diagnosis of lung cancer who met the inclusion criteria of the study and volunteered to participate in the study will constitute the sample of the study. 35 per group for the sample of the study. A total of 70 people will be sampled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Applications to the Intervention Group (Experimental): Patients with lung cancer admitted to the outpatient chemotherapy unit will be given pranayama breathing exercises every day for 4 weeks, covering 15-20 minutes. In patient education, the pranayama breathing exercise will be applied face-to-face by the researcher on the first day of chemotherapy treatment, before drug treatment. The application steps will be repeated until the patient learns, both by explaining and showing the patient, and if there are points that the patient cannot do, they will be corrected. When the patients are observed to perform the application fully and the chemotherapy treatments are finished, they will be asked to do the pranayama breathing exercise every day for 4 weeks, and with the same researcher 3 days a week (Monday, Wednesday, Saturday) with a smart phone whatsapp video call, the effectiveness and continuity of the application will be ensured and the patients will be monitored.
  Interventions: Procedure: Pranayama breathing exercise
- Applications to the Control Group (No Intervention): A pre-test will be applied to lung cancer patients in the control group who applied to the day chemotherapy unit. After the application of the personal information form and the quality of life scale, no breathing exercises will be performed. Individuals will continue their daily lives. After 4 weeks, the quality of life scale will be administered again. After the implementation of the quality of life scale, pranayama breathing exercise training will be given to all control group patients and they will be applied for 2 sessions.(The study will begin before the patients in both the experimental and control groups receive chemotherapy, which is their routine treatment).

INTERVENTIONS:
Procedure: Pranayama breathing exercise — Pranayama is an important step in yoga, way of life, and is translated as "the science of breathing, breath control, willful breathing". This alternating breathing-out action also balances the sympathetic and parasympathetic nervous systems, giving the person a state of calm, providing relaxation and positively affecting fatigue. Application steps; Right hand Nasika mudra is performed. Nasika mudra is the mudra where the second and third fingers of the right hand are folded into the palm and the other fingers are exposed. Then the right nostril is closed with the first finger of the right hand. Start by breathing through the left nostril. Then the left nostril is closed with the fourth finger and the breath is held. While the left nostril is closed, the right nostril is opened and inhaled. Breathe again through
  Arms: Applications to the Intervention Group

SUMMARY:
This research is a randomized controlled experimental study to determine the effect of pranayama breathing exercise applied to patients with lung cancer on quality of life.

DETAILED DESCRIPTION:
The population of the study consists of patients with primary diagnosis of lung cancer who applied to Erciyes University Health Practice and Research Center Nazende-Nuri Özkaya Oncology Day Treatment Center. Patients with primary diagnosis of lung cancer who met the inclusion criteria of the study and volunteered to participate in the study will constitute the sample of the study. It was calculated by performing power analysis for the sample of the study. In the power analysis made according to the effect size of the research; When calculating the partial eta square effect size of 0.06, alpha=0.05 and power=0.80 for two-way ANOVA in repeated measurements, the sample size per group is 35. A total of 70 people will be sampled. Data Collection Form and Tools: The data of the study are collected through Personal Information Form, European Cancer Research and Treatment Organization Quality of Life Scale 3rd Version, Informed Voluntary Consent Form, Eastern Cooperative Oncology Group (ECOG) Performance Scale, Mini Mental Test forms. The data of the research were obtained from the academic committee, ethics committee and institution of Erciyes University Faculty of Health Sciences. Patients who accept the study are pre-tested. Patient selection for the intervention and control groups of the study is made using the minimization randomization method. In the minimization method, the patients are assigned to groups according to age, gender, cancer cell type, cancer stage, duration and having a chronic disease. Data are collected from lung cancer patients who accepted to participate in the study, who applied to the outpatient chemotherapy unit by using face-to-face interview method by the researcher herself. During the study, the routine treatments of the patients in the intervention and control groups will not be interfered with.

Pre-Test: The patients with lung cancer who applied to the outpatient chemotherapy unit are informed about the research by the researcher and after obtaining the consent form, the personal information form and the quality of life scale are applied to the intervention and control groups by using the face-to-face interview method and the records obtained from the patient files, respectively.

Applications to the Intervention Group: Among the pranayama breathing exercises, only the Nadi Shothana technique will be applied to lung cancer patients who apply to the outpatient chemotherapy unit. This exercise will be done every day for 4 weeks, covering 15-20 minutes. After applying the personal information form and quality of life scale to the patients, the researcher will be informed about what the pranayama exercise is, its importance, purpose and benefits. Patients will be given an application guide and their questions will be answered if they have any. In patient education, the pranayama breathing exercise will be applied face-to-face by the researcher on the first day of chemotherapy treatment, before drug treatment. The application steps will be repeated until the patient learns, both by explaining and showing the patient, and if there are points that the patient cannot do, they will be corrected. When the patients are observed to perform the application fully and the chemotherapy treatments are finished, they will be asked to do the pranayama breathing exercise every day for 4 weeks, and with the same researcher 3 days a week (Monday, Wednesday, Saturday) with a smart phone whatsapp video call, the effectiveness and continuity of the application will be ensured and the patients will be monitored. If the patients assigned to the intervention group are unable to perform the application or have difficulties, the study with these patients will be terminated.

Applications to the Control Group: After the application of the personal information form and the quality of life scale, no breathing exercises will be performed. Individuals will continue their daily lives. After 4 weeks, the quality of life scale will be administered again. After the implementation of the quality of life scale, pranayama breathing exercise training will be given to all control group patients and they will be applied for 2 sessions.

Post-Test: The quality of life scale will be re-administered to the patients in both groups by the same researcher 4 weeks after the pre-test, and one day after the pranayama breathing exercise application to the control group and intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old,
2. Lung Cancer Stage III and IV,
3. Being literate,
4. Having sufficient communication skills,
5. Does not have any ailment that will reduce the ability to comprehend and understand,
6. Agreeing to participate in the research,
7. Knowing the diagnosis,
8. Receiving chemotherapy treatment,
9. ECOG performance score ≤ 2,
10. Not using opioids or sedating drugs,
11. Patients who can use smart phones themselves or their relatives will be included in the study

Exclusion Criteria:

1. Lung Cancer I., II., stage,
2. Receiving radiotherapy,
3. Having a history of Brain Metastasis,
4. Using integrated health practices in the treatment process,
5. Those who exercise regularly
6. For patients over 65 years of age, patients with a score below 24 on the mini mental test were not included in the study.

Research Termination Criteria

Intervention Group

1. Developing additional health problems,
2. Unwilling to continue the practice of pranayama breathing exercise,
3. Those who lost their lives during the research process,
4. Those who do not practice pranayama breathing exercise as recommended or cannot do it effectively,
5. The study will be terminated with patients who want to withdraw from the study.

Control Group

1. Developing additional health problems,
2. Those who lost their lives during the research process,
3. The study will be terminated with patients who want to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Quality of life of lung cancer patients | four weeks
  European Organization for Cancer Research and Treatment Quality of Life Scale :measure lung cancer patients before and four weeks aftter. European Organization for Cancer Research and Treatment Quality of Life Scale: scale consists of 3 sub-titles: general well-being, functional area and symptom control. While the maximum score that patients will get from these three sub-headings is 100, the minimum score is 0. The first 28 questions are questions related to the functional area and symptom control subheadings, and low scores on these questions mean high quality of life, and high scores mean low quality of life. The last two questions belong to the sub-heading of general well-being, and a low score on these questions indicates a low quality of life, and a high score indicates a high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We plan to share it after it is ready for publication.